CLINICAL TRIAL: NCT06653101
Title: Effect of Akkermansia Muciniphila Akk11 on Metabolic and Gut Health in Overweight and Obese Subjects: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effect of Akkermansia Muciniphila Akk11 on Metabolic and Gut Health in Overweight and Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2024014
Record Dates: First submitted 2024-10-16; First posted 2024-10-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-12

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Each Akk11 capsule contained 350 mg inulin and 175 mg FOS (2:1 ratio), together with 1 × 10¹⁰ AFU of viable Akk11 cells. Dosage: 3 capsules per day.
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Each placebo capsule contained 350 mg inulin and 175 mg FOS (2:1 ratio). Dosage: 3 capsules per day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The trial phase of this study lasted 8 weeks, and each patient will make 3 visits (week 0, week 4, week 8)
  Arms: Probiotic group
Dietary Supplement: Placebo — The trial phase of this study lasted 8 weeks, and each patient will make 3 visits (week 0, week 4, week 8)
  Arms: Placebo group

SUMMARY:
To assess the efficacy and safety of the use of probiotics as a food supplement compared to placebo in regulating body metabolism and gut microbiota in overweight or obese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. 18-45 years old;
2. BMI ≥ 24 kg/m2 or men with a body fat percentage of ≥ 25% and women with a body fat percentage of ≥ 30%；
3. Normal liver function indexes;
4. Willing to complete study-related questionnaires and diaries and complete all clinical visits.

Exclusion Criteria:

1. Those who have been diagnosed with high uric acid or gout are not recommended to participate in the test;
2. Psychiatric or neurological diseases, celiac disease, lactose intolerance, allergies;
3. Have the following diseases: irritable bowel syndrome, ulcerative colitis, fatty liver, liver cirrhosis, etc.;
4. Recently treated with antibiotics (i.e., < 3 months prior to the start of the study);
5. Participants who smoked more than 10 cigarettes per day were excluded;
6. It is not recommended to participate in other special circumstances, such as those who are allergic to probiotic products;
7. Pregnant and lactating women are not suitable for experiments.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Changes in serum concentrations of glucagon-like peptide-1 (GLP-1) before and after intervention. | week 0 and week 8
  Detected by enzyme-linked immunosorbent assay (ELISA).
Changes in serum concentrations of leptin before and after intervention. | week 0 and week 8
  Detected by enzyme-linked immunosorbent assay (ELISA).
Changes in serum concentrations of peptide YY before and after intervention. | week 0 and week 8
  Detected by enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Locations (1):
- Fei Xu, Zhengzhou, None Selected, China